CLINICAL TRIAL: NCT01137409
Title: Detecting Heart Disease Using First Pass Imaging With Gated SPECT Perfusion
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 0811004420
Record Dates: First submitted 2010-06-03; First posted 2010-06-04 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Suspected or Diagnosed with Coronary artery disease: All patients with suspected or previously diagnosed coronary artery disease

SUMMARY:
The aim of this study is to determine if stress first pass imaging in conjunction with a nuclear scan will improve the sensitivity for detecting heart disease. This study will also test the usefulness of a nuclear medicine camera, CDLCAM One Pass Angiography system.

DETAILED DESCRIPTION:
In this clinical trial, patients with suspected or previously diagnosed coronary artery disease who are clinically referred for either a treadmill exercise stress/rest SPECT study or a vasodilatation stress/rest SPECT study will be considered for this protocol. The vasodilation study may be either adenosine or regadenosin. In addition to the stress study, a stress/rest echocardiography study and first pass image will also be obtained. The reason to include echocardiography is to provide an independent measurement of the ejection fraction during pharmacological stress for comparison to the ejection fraction from the first pass study and from the ECG-gated SPECT study performed at rest. This will evaluate the added value of calculation of stress left ventricular ejection fraction (LVEF) over gated SPECT resting EF. This information will also assist in evaluating LV dysfunction following induction of pharmacological stress Nuclear imaging compared with echocardiographic stress EF, established imaging modalities for assessment of coronary heart disease.

The study will include two ECHO imaging sessions and two SPECT imaging sessions.

Patients will undergo a resting first pass image during the administration 99mTc-tetrofosmin; and a resting ECHO study at an appropriate imaging time. The resting ECHO will also be used to assess patient imaging window quality and to optimize equipment settings for subsequent stress images. A rest gated-SPECT image will be acquired at the appropriate imaging time.

The patient will then undergo a standard vasodilation stress infusion. A first pass image will be obtained during the administration of 99mTc-tetrofosmin. An ECHO will be obtained prior to the completion of the infusion. A gated-SPECT study will then be performed at the appropriate imaging time.

Tetrofosmin ECG-gated SPECT Imaging:

One hundred patients will be enrolled in the vasodilation stress/rest ECG-gated SPECT myocardial perfusion imaging group. Imaging time for each session will vary from one and a half to three hours. A one or two day imaging protocol can be utilized. Depending on what imaging session is done first (rest or stress), a "one-day" protocol consists of having the first dose of 99mTc-Tetrofosmin as a low dose of 10-15mCi. The second dose will be the high dose of 20-40mCi depending on the patient's weight. In the "two-day" protocol, patients will receive a high dose of 99mTc-Tetrofosmin for both imaging sessions. The dose given will depend on the patient's weight.

Rest Imaging:

If venous access is not already established, the standard universal precautions and 18-20 gauge catheter equipped with a 3-way stopcock will be inserted preferably in the antecubital vein. The patient will be injected with the appropriate amount of 99mTc-Tetrofosmin. The first pass image will be acquired during the injection (see first pass protocol). An Early resting gated-SPECT imaging and an ECHO will be done at 15 minutes and then repeated at 60 minutes (see ECHO protocol).

Adenosine Imaging:

If venous access is not already established, the standard universal precautions and 18-20 gauge catheter equipped with a 3-way stopcock will be inserted preferably in the antecubital vein. Patients will receive an infusion of adenosine at a rate of 140ug/kg/min. After 1.5 minutes of adenosine infusion, the appropriate dose of 99mTc-Tetrofosmin will be injected and adenosine infusion will continue for 4.5 additional minutes, in compliance with the standard 6-minute infusion protocol and current ASNC guidelines. The first pass image will be acquired during the injection (see first pass protocol). Blood pressure and heart rate will be documented every minute. 12 lead ECG will be obtained at baseline and printed once a minute. There will be continuous monitoring of ECG and symptoms throughout the infusion. The ECHO will be acquired at 2.5 min of adenosine infusion (see ECHO protocol). An Early resting gated-SPECT imaging and an ECHO will be done at 15 minutes post infusion and then repeated at 60 minutes.

Test Termination End Points (standard criteria)

* Symptomatic hypotension, bradycardia or high degree AV Block
* Severe shortness of breath or wheezing
* Completion of protocol
* ST Segment depression >2mm (horizontal or downsloping)
* Angina
* Life threatening arrhythmia
* Subject requests to stop

Regadenoson Imaging:

If venous access is not already established, the standard universal precautions and 18-20 gauge catheter equipped with a 3-way stopcock will be inserted preferably in the antecubital vein.

Patients will receive an infusion of Regadenoson (0.4 mg regadenoson) by rapid intravenous injection; followed immediately by 5 ml saline flush. 20-40 seconds after the saline flush Tetrofosmin is injected and a first pass image is done.

Patients will receive an infusion of Regadenoson at a rate of (0.4 mg regadenoson). After 1.5 minutes of Regadenoson infusion, the appropriate dose of 99mTc-Tetrofosmin will be injected and Regadenoson infusion will continue for 4.5 additional minutes, in compliance with the standard 6-minute infusion protocol and current ASNC guidelines. The first pass image will be acquired during the injection (see first pass protocol). Blood pressure and heart rate will be documented every minute. 12 lead ECG will be obtained at baseline and printed once a minute. There will be continuous monitoring of ECG and symptoms throughout the infusion. The ECHO will be acquired at 2.5 min of Regadenoson infusion (see ECHO protocol). An Early resting gated-SPECT imaging and an ECHO will be done at 15 minutes post infusion and then repeated at 60 minutes.

Test Termination End Points (standard criteria)

* Symptomatic hypotension, bradycardia or high degree AV Block
* Severe shortness of breath or wheezing
* Completion of protocol
* ST Segment depression >2mm (horizontal or downsloping)
* Angina
* Life threatening arrhythmia
* Subject requests to stop

Treadmill Exercise (Stress) Imaging:

If venous access is not already established, the standard universal precautions and 18-20 gauge catheter equipped with a 3-way stopcock will be inserted preferably in the antecubital vein. Patients will follow a preset treadmill protocol. ECG's will be continuously monitored during exercise and are printed out for each stage of exercise. Patients will be injected with the appropriate amount of 99mTc-Tetrofosmin. The first pass image will be acquired during the injection (see first pass protocol). Due to logistical difficulties, the ECHO will not be performed for this imaging session.

Test Termination End Points (standard criteria)

* Severe Fatigue
* ST segment depression or elevation >2mm (horizontal or downsloping)
* Severe Angina
* Severe Shortness of breath/ wheezing
* Significant drop (20mmHG) in blood pressure
* Significant elevation of blood pressure:
* Systolic :> 220mmHG
* Diastolic :> 120mmHG
* Severe lower extremity discomfort
* Signs of severe peripheral circulatory insufficiency: lightheadedness, nausea, pallor
* Onset of second or third degree AV Block
* Ventricular Tachycardia
* Symptomatic SVT
* Patient request to stop
* Completion of Protocol
* For a Nuclear Imaging Study, patient should reach 85% of age predicted maximum heart rate prior to the injection of radioisotope (220-age). Once target is reached then the isotope is injected and patient should exercise for 2 more minutes post injection

Echocardiography Imaging:

Instrument settings will be optimized to ensure the best delineation of the endocardial borders of the left ventricle. Rest ECHO will be obtained in the standard protocol for both imaging groups. Patients in the adenosine vasodilatation stress group will have an ECHO during the infusion of adenosine in the standard views. Patients in the exercise stress group will have an ECHO immediately after exercise in the standard views. Patients in both groups will have an ECHO 15 minutes and 60 minutes after stress.

2D and 3D- Echocardiography Views

Primary views:

* Apical four chamber 2D view (2D and color tissue Doppler)
* Apical two chamber 2D view (2D and color tissue Doppler)
* Apical 3D view

Secondary 2D views:

* Parasternal short axis at base, mid and apex of LV (2D and color tissue Doppler)
* Parasternal long axis

First Pass Radionuclide Angiography:

Patients are prepped as outlined previously including IV placement. For the resting image, patients are connected to the camera gate device for continuous registration of the ECG. Patients will be placed against the face of the camera to begin isotope infusion. The camera will detect the presence of the isotope within the SVC and initiate recording of the data; real time acquisition progress will be displayed on the computer screen.

During the acquisition for the treadmill exercise image, patients will be connected to the camera gate device for continuous registration of the ECG. Patients are placed against the face of the camera. The height of the camera is set to the patient and "Treadmill tracking" is set to the "ON" position. At peak exercise, the isotope is injected. The camera will detect the presence of the isotope within the SVC and initiate recording of the data; real time acquisition progress is displayed on the computer screen.

During acquisition for the adenosine vasodilatation image, patients are connected to the camera gate device for continuous registration of the ECG. Patients are placed against the face of the camera. The isotope is infused at 1.5 minutes of adenosine infusion. The camera will detect the presence of the isotope within the SVC and initiate recording of the data; real time acquisition progress is displayed on the computer screen.

The total image time for the first pass study is 30 seconds.

ELIGIBILITY:
Inclusion criteria:

* Males and females age 18 through 80 years
* Female patients who are: surgically sterile (hysterectomy or bilateral tubule libation), at least one year post-menopausal, or have a negative pregnancy test on the day of treatment
* Written informed consent

Exclusion Criteria:

* Patient consumed food/beverage/medication containing caffeine/methylxanthines up to 12 hours prior to infusion
* Exacerbation of COPD, Asthma (actively wheezing)
* Sinus node dysfunction in absence of pacemaker
* Use of Aggrenox (ASA/Dipyridamole), Pentoxifylline (Trental) , or oral Dipyridamole (Persantine)
* Atrial fibrillation
* Pregnant/breast feeding
* Non English speaking patients
* Subject is allergic or intolerant to aminophylline, regadenoson
* Subject has a history of known or suspected bronchospastic lung disease [e.g., asthma, wheezing, chronic obstructive pulmonary disease (COPD, etc.)]
* Patients with first degree or second degree AV block

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with suspected or previously diagnosed coronary artery disease that are clinically referred for either a treadmill exercise stress/rest SPECT study or an adenosine vasodilatation stress/rest SPECT study will be considered for this protocol. Efforts will be made to enroll equal numbers of men and women for this clinical study.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-08; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To determine if stress first pass imaging in conjunction with gated SPECT, with or with out low level exercise,will improve the sensitivity for detecting ischemic heart disease | First pass imaging done in conjunction with SPECT study
  First pass imaging will be done in conjunction with the clinically indicated SPECT study.

SECONDARY OUTCOMES:
To determine if first pass imaging provides a more reproducible approach for evaluation of both rest and stress global LV function over gated SPECT perfusion imaging compared with 3D echocardiography | Immediately following administration of regadenoson.
  Echocardiography will be done immediately following the administration of regadenoson.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Sinusas, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States